CLINICAL TRIAL: NCT03077685
Title: Phase IIa Trial Evaluating the Safety of Intratumoral Injection of NanoPac® in Subjects With Locally Advanced Pancreatic Adenocarcinoma
Brief Title: Trial of NanoPac® in Subjects With Locally Advanced Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NanOlogy, LLC (Industry)
Collaborators: US Biotest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NANOPAC-2016-05
Record Dates: First submitted 2017-02-28; First posted 2017-03-13 (Actual); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma
Keywords: pancreatic neoplasms; digestive system neoplasms; pancreatic diseases; digestive system diseases; pancreatic adenocarcinoma; pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Digestive System Neoplasms; Pancreatic Diseases; Digestive System Diseases | interventions — Paclitaxel

STUDY DESIGN:
Intervention Model Description: Open-label, dose-escalating, Phase IIa trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation: NanoPac® 6 mg/mL (Experimental): Intratumorally injected NanoPac® at a volume of up to 20% tumor volume
  Interventions: Drug: NanoPac®
- Dose Escalation: NanoPac® 10 mg/mL (Experimental): Intratumorally injected NanoPac® at a volume of up to 20% tumor volume
  Interventions: Drug: NanoPac®
- Dose Escalation: NanoPac® 15 mg/mL (Experimental): Intratumorally injected NanoPac® at a volume of up to 20% tumor volume
  Interventions: Drug: NanoPac®
- Second Phase: NanoPac® at Best Dose (Experimental): Intratumorally injected NanoPac® at a volume of up to 20% tumor volume. The dose administered in the second phase will be determined during the dose escalation phase. Subjects will receive two NanoPac® administrations, with the second injection administered one month after the first injection.
  Interventions: Drug: NanoPac®
- Third Phase: NanoPac® at Best Dose (Experimental): Intratumorally injected NanoPac® at a volume of up to 20% tumor volume. The dose administered in the third phase will be determined during the dose escalation phase. Subjects will receive four NanoPac® administrations, with the injections administered one month apart.
  Interventions: Drug: NanoPac®

INTERVENTIONS:
Drug: NanoPac® — Subjects with locally advanced pancreatic adenocarcinoma will receive intratumoral (ITU) NanoPac® (Sterile Nanoparticulate Paclitaxel) via endoscopic ultrasound-guided direct injection.
  Other Names: Paclitaxel

SUMMARY:
Open-label, dose-escalating, Phase IIa trial of NanoPac® to treat subjects with locally advanced pancreatic adenocarcinoma via direct intratumoral injection.

DETAILED DESCRIPTION:
In this open-label, dose-escalating, Phase IIa trial, subjects with locally advanced pancreatic adenocarcinoma will receive intratumoral (ITU) NanoPac® (Sterile Nanoparticulate Paclitaxel) via endoscopic ultrasound-guided direct injection.

Subjects will be enrolled in sequential cohorts of NanoPac® at escalating doses, at a volume based on up to 20% of calculated tumor volume (with a maximum injection volume of 5 mL per subject). During the first phase of the trial (dose escalation), each cohort will have three subjects, with cohorts enrolled sequentially starting at the lowest concentration. Following DSMB review of the cohort data, the next cohort may begin enrolling, an additional three subjects at the current dose may be enrolled, or if the first dose does not provide adequate safety and tolerability the study may be halted.

The dose determined to be most suitable for further evaluation, defined as the highest dose with an acceptable safety and tolerability profile as determined by the Data Safety Monitoring Board (DSMB), will be the dose used in the second phase of the study which will enroll 22 additional subjects who will receive two injections of NanoPac® at the same dose one month apart. In the third phase of the study, up to 30 subjects will receive up to four injections of NanoPac at the same dose, one month apart.

Plasma samples will be taken at various time points on the day of NanoPac® injection as well as once at each of the study visits, to characterize the pharmacokinetics (PK) of ITU NanoPac®.

Subjects will be followed for 12 months after NanoPac® injection for safety, overall survival (OS), progression-free survival (PFS), CA-19-9 levels, carcinoembryonic antigen (CEA) levels, reduction in pain, and tumor response to therapy (as shown by imaging).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Age ≥18 years;
* Histologically/cytologically confirmed locally advanced pancreatic adenocarcinoma; at least one lesion with a diameter of at least 1.5 cm but no more than 6 cm as documented via imaging (within 6 weeks of Screening);
* Subject not a candidate for surgery;
* Completion of at least one standard of care IV chemotherapy course for subjects in the dose escalation phase of the study. IV chemotherapy will be initiated prior to first NanoPac injection for subjects in the second and third phases. Hematologic recovery must be confirmed prior to study entry;
* Performance Status (ECOG) 0-1 at study entry;
* Life expectancy of at least 3 months;
* Adequate marrow, liver, and renal function at study entry:

  * ANC ≥ 1.5 x 109/L
  * Hemoglobin ≥ 9.5 grams/dL
  * Platelets ≥ 75 x 109/L
  * Total bilirubin ≤ 1.5x institutional ULN
  * AST/ ALT ≤ 2.5x institutional ULN
  * Creatinine ≤ 1.5x institutional ULN
* Effective contraception if the risk of conception exists.

Exclusion Criteria:

* Thrombotic or embolic events;
* Acute or subacute intestinal occlusion;
* History of inflammatory bowel disease;
* Known hypersensitivity to study drugs;
* Known drug or alcohol abuse;
* Pregnant or breastfeeding women;
* Previous or concurrent history of non-pancreatic malignancy except for non-melanoma skin cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shelagh Verco, PhD, Study Director — Vice President, Clinical Development, NanOlogy, LLC
Locations (4):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Parkview Cancer Institute, Fort Wayne, Indiana
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Taxol® (paclitaxel) Injection Package Insert. Bristol-Myers Squibb Company. Rev July 2011.
- [Background] ABRAXANE Package Insert. Celgene Company. Rev July 2015.
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Derived] Sharma NR, Lo SK, Hendifar A, Othman MO, Patel K, Mendoza-Ladd A, Verco S, Maulhardt HA, Verco J, Wendt A, Marin A, Schmidt CM, diZerega G. Response of Locally Advanced Pancreatic Cancer to Intratumoral Injection of Large Surface Area Microparticle Paclitaxel: Initial Report of Safety and Clinical Outcome. Pancreas. 2023 Mar 1;52(3):e179-e187. doi: 10.1097/MPA.0000000000002236. PMID 37782888

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Escalation: NanoPac® 6 mg/mL: Intratumorally injected NanoPac® 6 mg/mL at a volume of up to 20% tumor volume via endoscopic ultrasound-guided direct injection.
- Dose Escalation: NanoPac® 10 mg/mL: Intratumorally injected NanoPac® 10 mg/mL at a volume of up to 20% tumor volume via endoscopic ultrasound-guided direct injection.
- Dose Escalation: NanoPac® 15 mg/mL: Intratumorally injected NanoPac® 15 mg/mL at a volume of up to 20% tumor volume via endoscopic ultrasound-guided direct injection.
- Second Phase: NanoPac® 15 mg/mL: Intratumorally injected NanoPac® 15 mg/mL at a volume of up to 20% tumor volume via endoscopic ultrasound-guided direct injection. Subjects receive two NanoPac® administrations, with the second injection administered one month after the first injection.
- Third Phase: NanoPac® 15 mg/mL: Intratumorally injected NanoPac® 15 mg/mL at a volume of up to 20% tumor volume via endoscopic ultrasound-guided direct injection. Subjects receive up to four NanoPac® administrations, with injections administered one month apart.
Period: Overall Study
Arm/Group | Dose Escalation: NanoPac® 6 mg/mL | Dose Escalation: NanoPac® 10 mg/mL | Dose Escalation: NanoPac® 15 mg/mL | Second Phase: NanoPac® 15 mg/mL | Third Phase: NanoPac® 15 mg/mL
Started | 3 | 3 | 4 | 25 | 19
Completed | 2 | 3 | 2 | 19 | 8
Not Completed | 1 | 0 | 2 | 6 | 11
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 3
Not completed — Disease Progression | 1 | 0 | 0 | 2 | 1
Not completed — Withdrawn to proceed to surgery | 0 | 0 | 0 | 1 | 1
Not completed — Subject entered hospice care | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: NanoPac® 6 mg/mL | Dose Escalation: NanoPac® 10 mg/mL | Dose Escalation: NanoPac® 15 mg/mL | Second Phase: NanoPac® 15 mg/mL | Third Phase: NanoPac® 15 mg/mL | Total
Number analyzed (Participants) | 3 | 3 | 4 | 25 | 19 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (9.00) | 71.3 (8.08) | 72.0 (9.56) | 65.6 (10.08) | 71.3 (11.19) | 68.3 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 11 | 10 | 22
  Male | 2 | 3 | 4 | 14 | 9 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 4 | 7
  Not Hispanic or Latino | 2 | 2 | 3 | 25 | 15 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 4 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1 | 2
  White | 3 | 2 | 3 | 20 | 18 | 46
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 25 | 19 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events (Safety and Tolerability)
Description: Treatment Emergent Adverse Events will include laboratory assessments, physical examination findings, and vital signs.
Time Frame: Up to Week 24 for Dose Escalation subjects; up to Week 28 for Second Phase subjects; up to 9 Months for Third Phase subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: NanoPac® 6 mg/mL | Dose Escalation: NanoPac® 10 mg/mL | Dose Escalation: NanoPac® 15 mg/mL | Second Phase: NanoPac® 15 mg/mL | Third Phase: NanoPac® 15 mg/mL
Number analyzed (Participants) | 3 | 3 | 4 | 25 | 19
Participants
  Number of subjects with at least one TEAE | 3 | 3 | 4 | 23 | 19
  Number of subjects without any TEAE | 0 | 0 | 0 | 2 | 0

2. Secondary Outcome: Target Tumor Assessment
Description: Response was determined using RECIST 1.1 parameters (complete response, partial response, stable disease, progressive disease, unevaluable) for the treated lesion in all groups.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Groups:
- Second Phase: NanoPac® 15 mg/mL: Intratumorally injected NanoPac® 15 mg/mL at a volume of up to 20% tumor volume via endoscopic ultrasound-guided direct injection. Subjects received two NanoPac® administrations, with the second injection administered one month after the first injection.
- Third Phase: NanoPac® 15 mg/mL: Intratumorally injected NanoPac® 15 mg/mL at a volume of up to 20% tumor volume via endoscopic ultrasound-guided direct injection. Subjects received up to four NanoPac® administrations, with injections administered one month apart.
Arm/Group | Dose Escalation: NanoPac® 6 mg/mL | Dose Escalation: NanoPac® 10 mg/mL | Dose Escalation: NanoPac® 15 mg/mL | Second Phase: NanoPac® 15 mg/mL | Third Phase: NanoPac® 15 mg/mL
Number analyzed (Participants) | 3 | 3 | 4 | 25 | 19
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 1 | 0 | 2 | 3
  Stable Disease | 1 | 0 | 1 | 12 | 2
  Progressive Disease | 1 | 2 | 0 | 1 | 5
  Not evaluable | 1 | 0 | 3 | 10 | 9

3. Secondary Outcome: Plasma Paclitaxel Concentration (pg/mL)
Description: Plasma paclitaxel concentrations were analyzed in the dose escalation phase on Day 1 prior to injection and at 1, 2, 4, 6, and 24 hours after NanoPac injection, as well as at all other study visits. In the second and third phases, plasma paclitaxel concentrations were analyzed on Day 1 prior to NanoPac injection, and at 1 and 2 hours post NanoPac injection on all injection occasions, and at all study visits.
Time Frame: Day 1 and Week 24
Population: Not all subjects had data at all timepoints. On Day 1, data available for one subject in dose escalation 6 mg/mL, none in 10 mg/mL, and one in 15 mg/mL; second phase, six subjects; third phase three subjects. At Week 24, data available for one subject in dose escalation 6 mg/mL, none in 10 mg/mL, none in 15 mg/mL; second phase, eight subjects; third phase five subjects. Forty subjects received concomitant IV chemotherapy while on study; of these, 14 received concomitant taxane therapy.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Dose Escalation: NanoPac® 6 mg/mL | Dose Escalation: NanoPac® 10 mg/mL | Dose Escalation: NanoPac® 15 mg/mL | Second Phase: NanoPac® 15 mg/mL | Third Phase: NanoPac® 15 mg/mL
Number analyzed (Participants) | 2 | 0 | 1 | 11 | 7
pg/mL
  Day 1 Pre-Injection: number analyzed (Participants) | 1 | 0 | 1 | 6 | 3
  Day 1 Pre-Injection | 62.1 (NA) — Only 1 subject analyzed. |  | 304 (NA) — Only 1 subject analyzed. | 5497.0 (11887.04) | 17347.7 (27686.44)
  Week 24: number analyzed (Participants) | 1 | 0 | 0 | 8 | 5
  Week 24 | 30 (NA) — Only 1 subject analyzed. |  |  | 5017.8 (12139.23) | 63.2 (60.16)

4. Secondary Outcome: Pain (Visual Analog Scale) Score
Description: The visual analog scale (VAS) ranks pain from numbers 0 (no pain) to 10 (most pain). Lower scores mean a better outcome.
Time Frame: Day 1 (pre-injection) and Week 24
Population: Pain measured with VAS was not available for all subjects at all timepoints. For the Day 1 Pre-Injection timepoint, there was one subject in the 6 mg/mL dose escalation group for whom VAS was not available. For the Week 24 timepoint, there was one subject in the 6 mg/mL dose escalation group, three in the 15 mg/mL dose escalation group, 12 in the second phase, and 9 in the third phase for whom VAS data was not available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dose Escalation: NanoPac® 6 mg/mL | Dose Escalation: NanoPac® 10 mg/mL | Dose Escalation: NanoPac® 15 mg/mL | Second Phase: NanoPac® 15 mg/mL | Third Phase: NanoPac® 15 mg/mL
Number analyzed (Participants) | 2 | 3 | 4 | 25 | 19
units on a scale
  Day 1 (Pre-Injection) | 0 (0) | 0 (0) | 5.5 (4.12) | 1.2 (2.41) | 0.8 (1.42)
  Week 24: number analyzed (Participants) | 2 | 3 | 1 | 13 | 10
  Week 24 | 5.3 (3.18) | 0.8 (1.44) | 5.0 (NA) — Data only available from one subject | 1.7 (2.53) | 1.1 (2.23)

5. Secondary Outcome: Serum CA19-9 Level
Description: CA19-9 is a tumor marker for pancreatic cancer. Serum CA19-9 levels were assessed at all study visits.
Time Frame: Day 1 (Pre-Injection) and Week 24
Population: Missing CA19-9 data for Day 1: dose escalation 6 mg/mL two subjects; second phase two subjects; third phase three subjects. Missing CA19-9 data for Week 24: dose escalation 6 mg/mL one subject; dose escalation 15 mg/mL two subjects; second phase 10 subjects; third phase nine subjects.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Dose Escalation: NanoPac® 6 mg/mL | Dose Escalation: NanoPac® 10 mg/mL | Dose Escalation: NanoPac® 15 mg/mL | Second Phase: NanoPac® 15 mg/mL | Third Phase: NanoPac® 15 mg/mL
Number analyzed (Participants) | 2 | 3 | 4 | 25 | 19
U/mL
  Day 1 - Pre-Injection: number analyzed (Participants) | 1 | 3 | 4 | 23 | 16
  Day 1 - Pre-Injection | 248 (NA) — Data available for only one subject | 24 (24) | 2958 (4749) | 952 (2171) | 198 (362)
  Week 24: number analyzed (Participants) | 2 | 3 | 2 | 15 | 10
  Week 24 | 5476 (6396.49) | 49.3 (60.3) | 6179 (5402.3) | 141.6 (184.03) | 1222.6 (3126)

6. Secondary Outcome: Serum CEA Levels
Description: Carcinoembryonic antigen (CEA) is a tumor marker for pancreatic cancer.
Time Frame: Day 1 (Pre-Injection) and Week 24
Population: Missing CEA data for Day 1: dose escalation 6 mg/mL one subject; second phase two subjects; third phase two subjects. Missing CEA data for Week 24: dose escalation 6 mg/mL one subject; dose escalation 15 mg/mL three subjects; second phase 11 subjects; third phase nine subjects.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Dose Escalation: NanoPac® 6 mg/mL | Dose Escalation: NanoPac® 10 mg/mL | Dose Escalation: NanoPac® 15 mg/mL | Second Phase: NanoPac® 15 mg/mL | Third Phase: NanoPac® 15 mg/mL
Number analyzed (Participants) | 2 | 3 | 4 | 25 | 19
ug/L
  Day 1 - Pre-Injection: number analyzed (Participants) | 2 | 3 | 4 | 23 | 17
  Day 1 - Pre-Injection | 1.65 (0.778) | 27.1 (41.57) | 4.58 (1.68) | 5.17 (3.163) | 6.69 (5.976)
  Week 24: number analyzed (Participants) | 2 | 3 | 1 | 14 | 10
  Week 24 | 4.55 (2.758) | 53.33 (84.577) | 10.3 (NA) — Data available only for one subject | 5.49 (3.291) | 13.04 (16.718)

ADVERSE EVENTS:
Time Frame: Up to 9 months
Description: AEs were collected at all study visits from the time of dosing. Subjects were required to spontaneously report any AE. Study personnel asked open-ended questions to obtain information about AEs at every visit. Total AEs are reported in this record regardless of relationship to study treatment.
Arm/Group | Dose Escalation: NanoPac® 6 mg/mL | Dose Escalation: NanoPac® 10 mg/mL | Dose Escalation: NanoPac® 15 mg/mL | Second Phase: NanoPac® 15 mg/mL | Third Phase: NanoPac® 15 mg/mL
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/4 | 1/25 | 3/19
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 3/4 | 13/25 | 8/19
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 23/25 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: NanoPac® 6 mg/mL (N=3) | Dose Escalation: NanoPac® 10 mg/mL (N=3) | Dose Escalation: NanoPac® 15 mg/mL (N=4) | Second Phase: NanoPac® 15 mg/mL (N=25) | Third Phase: NanoPac® 15 mg/mL (N=19)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (4) | 2 (2) | 1 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 3 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation: NanoPac® 6 mg/mL (N=3) | Dose Escalation: NanoPac® 10 mg/mL (N=3) | Dose Escalation: NanoPac® 15 mg/mL (N=4) | Second Phase: NanoPac® 15 mg/mL (N=25) | Third Phase: NanoPac® 15 mg/mL (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 10 (16) | 6 (7)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 7 (8) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (8) | 2 (4)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 9 (9) | 6 (11)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (2)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Full blood count abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic enzymes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 6 (7) | 3 (4)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 5 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Senile osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder trabeculation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Choluria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Antiviral prophylaxis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/85/NCT03077685/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT03077685/SAP_001.pdf